CLINICAL TRIAL: NCT04430361
Title: Comparison of the Efficacy and Safety of 5-HT3 Receptor Antagonist, Dexamethasone or Megestrol Acetate Dispersible Tablets in the Control of Nausea and Vomiting Induced by Highly Emetogenic Chemotherapy: a Prospective, Randomized Controlled Phase II Clinical Trial
Brief Title: the Efficacy and Safety of 5-HT3 Receptor Antagonist, Dexamethasone or Megestrol Acetate Dispersible Tablets in the Control of Nausea and Vomiting Induced by Highly Emetogenic Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017098
Record Dates: First submitted 2020-05-26; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-05

CONDITIONS: Tumor; Chemotherapy-induced Nausea and Vomiting
Keywords: Megestrol; Tumor; Cisplatin; Chemotherapy-induced nausea and vomiting; Highly emetogenic chemotherapy
MeSH Terms: conditions — Neoplasms; Vomiting | interventions — Megestrol; Megestrol Acetate; Serotonin 5-HT3 Receptor Antagonists; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Megestrol (Experimental): Palonosetron 2.5mg, Dexamethasone 12mg on the first day, 8mg on the 2nd-4th day, Megestrol acetates 160mg orally every morning on the day of the beginning of chemotherapy for 10 days.
  Interventions: Drug: Megestrol; Drug: 5-HT3 receptor antagonist; Drug: dexamethasone
- Control (Other): Palonosetron 2.5mg, Dexamethasone12mg on the first day, 8mg on the 2nd-4th day
  Interventions: Drug: 5-HT3 receptor antagonist; Drug: dexamethasone

INTERVENTIONS:
Drug: Megestrol — 160 mg of megestrol acetate dispersible tablets were taken orally every morning on the day of the beginning of chemotherapy for 10 days.
  Other Names: Megestrol acetate
  Arms: Megestrol
Drug: 5-HT3 receptor antagonist — 5-HT3 receptor antagonist 2.5mg/iv
Drug: dexamethasone — dexamethasone 12mg on the first day, 8mg on the 2nd-4th day,

SUMMARY:
To compare the efficacy and safety of megestrol acetate dispersible tablets combined with 5-HT3 receptor antagonist and dexamethasone triple antiemetic regimen and 5-HT3 receptor antagonist and dexamethasone combined antiemetic regimen in the control of CINV induced by hyperemetic chemotherapy.

DETAILED DESCRIPTION:
120 patients with malignant tumors diagnosed by pathology or cytology and treated with highly emetogenic chemotherapy drugs containing cisplatin from September 2018 to December 2019 were selected. The patients were randomly assigned to megestrol group (megestrol acetate dispersible tablets+5-HT3 receptor antagonist+dexamethasone) or control group (5-HT3 receptor antagonist + dexamethasone) at 1:1. The dosage of antiemetic drugs in the control group: 5-HT3 receptor antagonist 2.5mg, dexamethasone 12mg on the first day, 8mg on the 2nd-4th day, all were injected intravenously with 30min before chemotherapy for 5 days. The patients in the megestrol acetate group were given megestrol acetate dispersible tablets on the basis of the control group. 160 mg of megestrol acetate dispersible tablets were taken orally every morning on the day of the beginning of chemotherapy for 10 days. The main end point was the proportion of control of nausea and vomiting between the two groups during the delayed period (24-120 hours after the beginning of chemotherapy), that is, the proportion of complete remission (no vomiting and no need for rescue treatment) and complete prevention (no nausea and vomiting).The secondary end point was the control ratio of nausea and vomiting in the acute phase (0-24 hours after the beginning of chemotherapy) and the overall phase (0-120 hours after the beginning of chemotherapy); the proportion of patients with grade 3-4 nausea and vomiting during chemotherapy; the adverse reactions related to antiemetic drugs and the score of quality of life of patients in both groups before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Tumor patients diagnosed by histopathology or cytology, as long as the chemotherapy with cisplatin is used, the amount of cisplatin is 60-80 mg/m2;
* Unlimited gender, age 18 to 70 years old;
* ECOG physical status score 0-1;
* The survival time is predicted to be more than 3 months;
* Bone marrow hematopoietic function was not significantly impaired (WBC≥3.5109/L, ANC≥1.5109/L, PLT≥100109/L, Hb≥100g/L);
* Biochemical examination AST / ALT ≤ 2.5 times the upper limit of normal; bilirubin ≤ 1.5 times the upper limit of normal; creatinine clearance ≥ 60ml / min, normal ECG;
* Signing informed consent;

Exclusion Criteria:

* Women who are pregnant or breastfeeding, women of childbearing age who refuse to receive contraception;
* Brain metastasis;
* Combine all of the following serious or uncontrolled diseases that affect participation in the trial: Uncontrollable hypertension, history of unstable hypertension, or poor adherence to antihypertention drugs; Unstable angina; Symptomatic congestive heart failure; Myocardial infarction occurred within 6 months before enrollment; Severe uncontrollable arrhythmia; Uncontrollable diabetes; Active or uncontrollable infection; Intestinal paralysis, intestinal obstruction, interstitial pneumonia, active gastric ulcer; Subject to immunosuppressive therapy;
* Inability to understand or express informed consent;
* The investigator judged other conditions that were not suitable for clinical research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-09-07 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of control of nausea and vomiting between the two groups during the delayed period | 24 to120 hours
  The main end point was the proportion of control of nausea and vomiting between the two groups during the delayed period chemotherapy

SECONDARY OUTCOMES:
The control ratio of nausea and vomiting in the acute phase and the overall phase | 0 to 120 hours
  The control ratio of nausea and vomiting in the acute phase and the overall phase
The proportion of patients with grade 3-4 vomiting | 0 to 120 hours
  The proportion of patients with grade 3-4 vomiting during chemotherapy
The adverse reactions related to antiemetic drugs | 1 mounth
  The adverse reactions related to antiemetic drugs of patients in both groups before and after treatment.
The score of quality of life of patients | 1 mounth
  The score of quality of life of patients in both groups before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, Principal Investigator — Henan Cancer Hospital; Ning Li, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No